CLINICAL TRIAL: NCT05179824
Title: Tempus Priority Study: An Observational Study of Patients Who Have Received Comprehensive Genomic Profiling
Brief Title: Tempus Priority Study: A Pan-tumor Observational Study
Status: Active, not recruiting | Type: Observational
Sponsor: Tempus AI (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CA-001
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Prostate Cancer; Bladder Cancer; Lung Cancer; Brain Cancer; Pancreatic Cancer; Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Cancer of Liver; Cancer of Colon; Cancer of Head and Neck; Cancer of Stomach; Cancer of Gastrointestinal Tract; Cancer of Rectum; Cancer of Esophagus; Cancer of Skin; Cancer of Cervix; Cancer of Kidney; Cancer of Larynx; Cancer of Endometrium; Cancer of the Bile Duct; Cancer of Vulva; Cancer of Bone and Connective Tissue; Leukemia; Lymphoma; Spinal Cord Cancer
Keywords: Cancer; Oncology; Observational; Genomic Profiling; Precision Medicine
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms; Lung Neoplasms; Brain Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Liver Neoplasms; Colonic Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Gastrointestinal Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Skin Neoplasms; Uterine Cervical Neoplasms; Kidney Neoplasms; Laryngeal Neoplasms; Endometrial Neoplasms; Bile Duct Neoplasms; Vulvar Neoplasms; Bone Neoplasms; Leukemia; Lymphoma; Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Archival tissue will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: Standard of Care (SOC) CGP: This group will facilitate collection of paired clinical and molecular data done as part of the standard of care or routine clinical care across a variety of institutions. The goal of Group 1 is to capture a broad range of participants to better understand longitudinal outcomes across institutions and standards of care.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No Intervention

SUMMARY:
Observational study that will be collecting clinical and molecular health information from cancer patients who have received comprehensive genomic profiling and meet the specific eligibility criteria outlined for each cohort with the goal of conducting research to advance cancer care and create a dataset that furthers cancer research.

DETAILED DESCRIPTION:
The Study will collect combined clinical and molecular health information for cancer patients in the United States from multiple academic medical centers and community oncology practices. Participants who agree to join the Study will have their molecular profiling results, associated clinical health information, and longitudinal outcomes health information collected by the participating Institution for submission to Tempus. The specific goal of the Study is to create an outcomes-based dataset for future research to improve cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Solid or hematologic malignancy.
2. Willing and able to provide informed consent where required.
3. Has received or will receive genomic profiling.

Exclusion Criteria:

1. Individuals without the capacity to consent.
2. Prisoners at the time of enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This protocol targets a broad spectrum of cancer patients with comprehensive genomic profiling.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2030-10-19 (Estimated)

PRIMARY OUTCOMES:
Create robust data set of health information | Up to 10 years
  To create a robust data set of health information about cancer patients who receive comprehensive genomic profiling in order to facilitate future novel precision medicine research

SECONDARY OUTCOMES:
Document clinical events for patients who have had comprehensive genomic profiling | Up to 10 years
  To document specific clinical events in relation to diagnosis, treatment, and outcomes for patients who have had comprehensive genomic profiling
Evaluate longitudinal paired tissue and cell free molecular testing | Up to 10 years
  To evaluate the feasibility of longitudinal paired tissue and cell free molecular testing of participants with specific types of cancer, mutations, or therapies

OTHER OUTCOMES:
Support prospective and retrospective research studies | Up to 10 years
  To support prospective and retrospective research studies on participants with specific cancer types
Describe real world treatment outcomes | Up to 10 years
  To describe real world treatment outcomes (such as real-world response, real world duration of response, real world progression free survival, real world time to next treatment, real world time to treatment discontinuation, and overall survival)
Review medical information for standard of care decisions and health outcomes | Up to 10 years
  To review medical information for standard of care decisions in the future and general health outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Kristiyana Kaneva, MD, MS, MBA, Principal Investigator — Tempus AI, Inc.
Locations (2):
- United States (2):
  - UT Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zehir A, Benayed R, Shah RH, Syed A, Middha S, Kim HR, Srinivasan P, Gao J, Chakravarty D, Devlin SM, Hellmann MD, Barron DA, Schram AM, Hameed M, Dogan S, Ross DS, Hechtman JF, DeLair DF, Yao J, Mandelker DL, Cheng DT, Chandramohan R, Mohanty AS, Ptashkin RN, Jayakumaran G, Prasad M, Syed MH, Rema AB, Liu ZY, Nafa K, Borsu L, Sadowska J, Casanova J, Bacares R, Kiecka IJ, Razumova A, Son JB, Stewart L, Baldi T, Mullaney KA, Al-Ahmadie H, Vakiani E, Abeshouse AA, Penson AV, Jonsson P, Camacho N, Chang MT, Won HH, Gross BE, Kundra R, Heins ZJ, Chen HW, Phillips S, Zhang H, Wang J, Ochoa A, Wills J, Eubank M, Thomas SB, Gardos SM, Reales DN, Galle J, Durany R, Cambria R, Abida W, Cercek A, Feldman DR, Gounder MM, Hakimi AA, Harding JJ, Iyer G, Janjigian YY, Jordan EJ, Kelly CM, Lowery MA, Morris LGT, Omuro AM, Raj N, Razavi P, Shoushtari AN, Shukla N, Soumerai TE, Varghese AM, Yaeger R, Coleman J, Bochner B, Riely GJ, Saltz LB, Scher HI, Sabbatini PJ, Robson ME, Klimstra DS, Taylor BS, Baselga J, Schultz N, Hyman DM, Arcila ME, Solit DB, Ladanyi M, Berger MF. Mutational landscape of metastatic cancer revealed from prospective clinical sequencing of 10,000 patients. Nat Med. 2017 Jun;23(6):703-713. doi: 10.1038/nm.4333. Epub 2017 May 8. PMID 28481359
- [Background] Daoud A, Chu QS. Targeting Novel but Less Common Driver Mutations and Chromosomal Translocations in Advanced Non-Small Cell Lung Cancer. Front Oncol. 2017 Sep 29;7:222. doi: 10.3389/fonc.2017.00222. eCollection 2017. PMID 29034207
- [Background] Ersek JL, Black LJ, Thompson MA, Kim ES. Implementing Precision Medicine Programs and Clinical Trials in the Community-Based Oncology Practice: Barriers and Best Practices. Am Soc Clin Oncol Educ Book. 2018 May 23;38:188-196. doi: 10.1200/EDBK_200633. PMID 30231363
- [Background] Griffith SD, Tucker M, Bowser B, Calkins G, Chang CJ, Guardino E, Khozin S, Kraut J, You P, Schrag D, Miksad RA. Generating Real-World Tumor Burden Endpoints from Electronic Health Record Data: Comparison of RECIST, Radiology-Anchored, and Clinician-Anchored Approaches for Abstracting Real-World Progression in Non-Small Cell Lung Cancer. Adv Ther. 2019 Aug;36(8):2122-2136. doi: 10.1007/s12325-019-00970-1. Epub 2019 May 28. PMID 31140124